CLINICAL TRIAL: NCT07386509
Title: WU 345: Immune Responses to Adjuvanted and Non-adjuvanted Seasonal Influenza
Brief Title: WU 345: Immune Responses to Adjuvanted and Non-adjuvanted Seasonal Influenza Vaccines in the Lymphoid Tissues.
Acronym: WU 345
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: COVID pandemic No participant experiences (benefits, adverse events/adverse reactions)to report. There have been no safety concerns in either participant.
  No minor deviations to report
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 201912144
Record Dates: First submitted 2026-01-27; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Healthy
Keywords: immunue response

STUDY DESIGN:
Intervention Model Description: All subjects will concomitantly receive a single dose of both Fluad® and Afluria® administered intramuscularly in opposite deltoid muscles.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single dose of both Fluad® and Afluria® (Experimental): All subjects will concomitantly receive a single dose of both Fluad® and Afluria® administered intramuscularly
  Interventions: Drug: Fluad® and Afluria® vaccination

INTERVENTIONS:
Drug: Fluad® and Afluria® vaccination — All subjects will concomitantly receive a single dose of both Fluad® and Afluria® administered intramuscularly in opposite deltoid muscles

SUMMARY:
Healthy adults (18-49 years of age) with no previous influenza virus vaccination history for at least three years prior to enrollment will be recruited to participate in this study. All subjects will concomitantly receive a single dose of both Fluad® and Afluria® administered intramuscularly in opposite deltoid muscles. Blood samples collected at 9 visits (screening, baseline, days 7, 14, 28, 60, 90, 120 and 180, fine needle aspiration (FNAs) from axillary lymph nodes from both axillae at baseline, days 7, 14, 28, 60, 90, 120 and 180.

DETAILED DESCRIPTION:
Healthy adults (18-49 years of age) with no previous influenza virus vaccination history for at least three years prior to enrollment will be recruited to participate in this study. All subjects will concomitantly receive a single dose of both Fluad® and Afluria® administered intramuscularly in opposite deltoid muscles. Blood samples collected at 9 visits (screening, baseline, days 7, 14, 28, 60, 90, 120 and 180, fine needle aspiration (FNAs) from axillary lymph nodes from both axillae at baseline, days 7, 14, 28, 60, 90, 120 and 180.

ELIGIBILITY:
Inclusion Criteria:

* 1. Healthy subjects aged 18-49 years. 2. Able to understand and give informed consent. 3. Women of child-bearing potential (not surgically sterile via tubal ligation, bilateral oophorectomy or hysterectomy or who are not postmenopausal for ≥1 year) must agree to practice adequate contraception that may include, but is not limited to, abstinence, monogamous relationship with vasectomized partner, barrier methods such as condoms, diaphragms, spermicides, intrauterine devices, and licensed hormonal methods* for 28 days before and 28 days after rabies vaccination.

  * Women of child-bearing potential using licensed hormonal methods must also use a second form of contraception.

    4. Are in good health, as determined by medical history and targeted physical exam related to this history.

    5. Willing to give FNA specimens for the study.

    6. The following laboratory values obtained within 14 days prior to entry by any US laboratory that has a CLIA certification or its equivalent.

    • Absolute neutrophil count (ANC) ≥750 cells/mm3

    • Hemoglobin ≥11.0 g/dL for men and ≥10.0 g/dL for women
    * Platelet count ≥100,000/mm3
    * Creatinine clearance ≥60 mL/min estimated by the Cockcroft-Gault equation
    * NOTE: A program for calculating creatinine clearance by the Cockcroft-Gault method is available on www.fstrf.org
    * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) (SGPT) ≤5.0 times upper limit of normal (ULN)
    * Erythrocyte sedimentation rate (ESR) within normal range

Exclusion Criteria:

* 1. Receipt of the following:

  * Receipt of blood products 3 months prior to vaccination or expected receipt through 12 months after vaccination.
  * Receipt of any live virus vaccines within 28 days prior to vaccination or expected receipt within 28 days after vaccination. *
  * Receipt of any inactivated vaccine within 14 days or expected receipt within 14 days after vaccination other than study vaccine. * 2. Presence of co-morbidities or immunosuppressive states such as: Chronic medical problems including (but not limited to) insulin dependent diabetes, severe heart disease (including arrhythmias), severe lung disease, auto immune diseases, thrombocytopenia and any other severe medical conditions.

    3. Alcohol abuse, drug abuse, or psychiatric conditions that in the opinion of the investigator would preclude compliance with the trial or interpretation of safety or endpoint data.

    4. Any history of lymphoma involving axillary nodes or any history of breast cancer.

    5. Impaired immune function or known chronic infections including, but not limited to, known HIV, tuberculosis, hepatitis B or C; organ transplantation (bone marrow, hematopoietic stem cell, or solid organ transplant); immunosuppression due to cancer; current and/or expected receipt of chemotherapy, radiation therapy, steroids** (i.e., more than 20 mg of prednisone given daily or on alternative days for 2 weeks or more in the past 90 days , or high dose inhaled corticosteroids***); and any other immunosuppressive therapies (including anti-TNF therapy), functional or anatomic asplenia, or congenital immunodeficiency.

    6. Pregnancy or breast feeding 7. Conditions that could affect the safety of the volunteers, such as:
  * Severe reactions to prior vaccinations, including anaphylaxis
  * History of Guillain-Barré syndrome
  * History of bleeding disorders or current use of warfarin, aspirin, heparin, nonsteroidal anti-inflammatory drugs (NSAIDs) or other blood thinner/anticoagulant medications in the past week
  * Any allergy to any component of the vaccine or lidocaine 8. Subjects with any acute illness, including any fever (> 100.4 F [>38.0C], regardless of the route) within 3 days prior to vaccination *.

    9. Social, occupational, or any other condition that in the opinion of the investigator might interfere with compliance with the study and vaccine evaluation.

    10. ESR>30 mm/hour. 11. Previously received the 2019-2020 influenza vaccine. 12. Bilateral inflammatory process of upper arms in the past 2 weeks. 13. Prior breast or axillary biopsy and/or surgery.

Notes:

* An individual who initially is excluded from study participation based on one or more of the time-limited exclusion criteria (e.g., acute illness, receipt or expected receipt of live or inactivated vaccines) may be reconsidered for enrollment once the condition has resolved as long as the subject continues to meet all other entry criteria.

  * Subjects receiving > 20 mg/day of prednisone or its equivalent daily or on alternate days for more than 2 weeks may enter the study after therapy has been discontinued for more than 3 months.

    * Subjects are excluded if on high dose intranasal steroids defined as > 960 mcg/day of beclomethasone dipropionate or equivalent.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2020-03-17 (Actual); Primary Completion 2022-11-04 (Actual); Study Completion 2022-11-04 (Actual)

PRIMARY OUTCOMES:
Comparison of antibody titers at Day 28 versus baseline | Baseline and Day 28

SECONDARY OUTCOMES:
Frequency, severity, and causality of all adverse events. | Baseline and Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Presti, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine Infectious Disease Clinical Trials Unit., St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Informed Consent Form (2021-12-07): https://cdn.clinicaltrials.gov/large-docs/09/NCT07386509/ICF_000.pdf